CLINICAL TRIAL: NCT02408315
Title: Induction With Misoprostol: Oral Mucosa Versus Vaginal Epithelium
Brief Title: Induction With Misoprostol: Oral Mucosa Versus Vaginal Epithelium (IMPROVE)
Acronym: IMPROVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, David Haas, Professor Vice Chair for Research, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: IMPROVE
Record Dates: First submitted 2015-02-10; First posted 2015-04-03 (Estimated); Results first posted 2019-07-09 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-03

CONDITIONS: Pregnancy
Keywords: induction of labor; safety; pharmacokinetic; misoprostol
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- misoprostol/placebo using buccal (Placebo Comparator): Randomized for buccal route of administration/ placebo
  Interventions: Drug: misoprostol/placebo
- misoprostol/placebo using vaginal (Placebo Comparator): Randomized for vaginal route of administration/ placebo
  Interventions: Drug: misoprostol/placebo

INTERVENTIONS:
Drug: misoprostol/placebo — buccal or vaginal routes of administration/ placebo to compare methods for efficacy and safety during induction.
  Other Names: Cytotec

SUMMARY:
The primary objective of this study is to compare the efficacy and safety of vaginal and buccal misoprostol for women undergoing labor induction at greater than or equal to 37+ 0 completed weeks gestation. Thus, the investigators have both efficacy and a safety primary outcomes.

The secondary objective of this study is to assess the pharmacokinetic(PK) parameters with these two routes of administration in a sub-cohort of this trial. The long term objective of this line of research is to inform providers' clinical decision making for the large number of women having labor induction. By providing robust PK and pharmacodynamic (PD) evaluation, clinical outcomes data for these two routes of administration, clinicians will be informed for evidence-based decisions about the preferred route of administration of misoprostol.

DETAILED DESCRIPTION:
Misoprostol is currently administered in many different ways. It can be administered vaginally, rectally, orally, buccally, and sublingually. Each route has its benefits and potential drawbacks. While vaginal administration is most common, recent trends in practice have yielded more buccal use of this drug. There is extensive clinical experience with this agent and a large body of published reports supporting its safety and efficacy when used appropriately. However, we only found one published trial directly comparing buccal to vaginal misoprostol head-to-head. In that trial, there were no significant differences in any of the outcomes other than higher rates of tachysystole in the buccal group. However, this trial utilized higher doses of misoprostol (up to 100mcg) than are typically used clinically per the ACOG Practice Bulletin (starting at 25 mcg).

Additionally, there are few comparisons of the pharmacokinetics of misoprostol between the buccal and vaginal routes. In fact, all of the PK studies comparing these routes are in women undergoing pregnancy terminations in the 1st or 2nd trimesters and do not include women undergoing labor induction at term. As the physiological changes in pregnancy have a profound impact on drug metabolism and disposition, this is an important gap in the current knowledge.

The 3 Specific Aims of this trial are:

1. To compare the efficacy and safety of 25 mcg of misoprostol initially followed by 50mcg thereafter administered by either buccal or vaginal route in a placebo-controlled, double blind RCT. We will recruit women at term undergoing labor induction to accomplish this trial.
2. To compare the PK parameters of 25 mcg and 50 mcg of misoprostol administered by either buccal or vaginal routes. Further, we will analyze the clinical outcomes in Aim 1 based on the PK parameters, controlling for patient characteristics, to assess the impact of PK parameters on clinical success of this drug. In this way, we hope to comment on the strategic dose and individualized dosing model potential for labor induction with misoprostol.
3. To compare the trial participant satisfaction with each route of administration to improve patient-based outcomes. This will be done by administering a satisfaction survey at the end of the trial. As participants will have study drug placed both buccally and vaginally, they will be uniquely able to comment on comfort and preference for route of delivery.

We will recruit women who are admitted for term labor induction and for whom the provider plans to utilize misoprostol. Women will be randomized to receive either buccal or vaginal misoprostol; first dose will be 25 mcg followed by 50mcg for subsequent doses. Three hundred women will be recruited to the overall trial and a subcohort of 60 women will be recruited to participate in the PK portion of the trial.

ELIGIBILITY:
Inclusion Criteria:

* A medical indication for induction of labor at a gestational age between 37 +0 and 38 +6 weeks OR an elective or medical indication for induction of labor at a gestational age greater than or equal to 39 + 0 completed weeks
* Participant age of greater than or equal to14 years old
* Singleton pregnancy
* Modified Bishop score of less than or equal to 6
* Vertex fetal presentation by examination or ultrasound
* Any membrane status

Exclusion Criteria:

* Elective inductions between 37 +0 and 38 +6 completed weeks are specifically excluded
* Known intrauterine fetal demise
* Any uterine scar including prior cesarean section and myomectomy
* Known major fetal congenital malformations that may impact neonatal health
* Other evidence of fetal compromise (such as Category 2 or 3 tracing) before the induction begins
* Prior induction/cervical ripening methods utilized during this pregnancy
* Allergy to misoprostol
* Known untreated cervical infection (e.g. Gonorrhea, Chlamydia)
* Planned cesarean section due to maternal or fetal condition
* Any other contraindication to labor induction or misoprostol therapy

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2015-09; Primary Completion 2017-11 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Haas, MD, Principal Investigator — IU School of Medicine
Locations (2):
- United States (2):
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: Yes
Will share as needed for IPD.
Supporting Information: Study Protocol, ICF
Time Frame: After study completion and for 1 year after
Access Criteria: Email contact to study contact.

REFERENCES:
- [Background] Nassar AH, Awwad J, Khalil AM, Abu-Musa A, Mehio G, Usta IM. A randomised comparison of patient satisfaction with vaginal and sublingual misoprostol for induction of labour at term. BJOG. 2007 Oct;114(10):1215-21. doi: 10.1111/j.1471-0528.2007.01492.x. PMID 17877674
- [Derived] Vorontsova Y, Haas DM, Flannery K, Masters AR, Silva LL, Pierson RC, Yeley B, Hogg G, Guise D, Heathman M, Quinney SK. Pharmacokinetics of vaginal versus buccal misoprostol for labor induction at term. Clin Transl Sci. 2022 Aug;15(8):1937-1945. doi: 10.1111/cts.13306. Epub 2022 Jun 12. PMID 35587540
- [Derived] Haas DM, Daggy J, Flannery KM, Dorr ML, Bonsack C, Bhamidipalli SS, Pierson RC, Lathrop A, Towns R, Ngo N, Head A, Morgan S, Quinney SK. A comparison of vaginal versus buccal misoprostol for cervical ripening in women for labor induction at term (the IMPROVE trial): a triple-masked randomized controlled trial. Am J Obstet Gynecol. 2019 Sep;221(3):259.e1-259.e16. doi: 10.1016/j.ajog.2019.04.037. Epub 2019 May 7. PMID 31075246

RESULTS

PARTICIPANT FLOW:
Groups:
- Buccal Misoprostol/Vaginal Placebo: Misoprostol administered buccally with placebo administered vaginally.
- Vaginal Misoprostol/Buccal Placebo: Misoprostol administered vaginally with placebo administered buccally.
Period: Overall Study
Arm/Group | Buccal Misoprostol/Vaginal Placebo | Vaginal Misoprostol/Buccal Placebo
Started | 148 | 152
Completed | 148 | 152
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buccal Misoprostol/Vaginal Placebo | Vaginal Misoprostol/Buccal Placebo | Total
Number analyzed (Participants) | 148 | 152 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 4
  Between 18 and 65 years | 146 | 150 | 296
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.59 (6.4) | 28.21 (6.4) | 27.91 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 152 | 300
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 49 | 45 | 94
  White | 66 | 74 | 140
  More than one race | 5 | 3 | 8
  Unknown or Not Reported | 27 | 29 | 56
Region of Enrollment [Number; unit: participants]
  United States | 148 | 152 | 300

OUTCOME MEASURES:

1. Primary Outcome: Time to Delivery
Description: number of hours from placement of study drug to delivery
  Cesarean delivery for fetal non--reassurance indication
Time Frame: from study entry until delivery- anticipated 3 days
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Buccal Misoprostol/Vaginal Placebo | Vaginal Misoprostol/Buccal Placebo
Number analyzed (Participants) | 148 | 152
hours | 28.1 [24.1 to 31.4] | 20.1 [18.2 to 22.8]
Statistical Analysis 1: Comparison: Buccal Misoprostol/Vaginal Placebo vs Vaginal Misoprostol/Buccal Placebo; Test type: Non-Inferiority — Estimates obtained from Kaplan-Meier method and results of Log-rank test. P-value for non-inferiority hypothesis based on Cox proportional hazards model (H0: HR ≤ 0.74 vs. HA: HR > .74), p-value < .05 provides evidence to reject inferiority and conclude BM is non-inferior to VM; p = 0.663, Cox proportional

2. Primary Outcome: Number of Participants With Cesarean Deliveries Based on Fetal Non-Reassurance Indications
Description: Rate of cesarean deliveries performed for fetal non-reassurance as the indication
Time Frame: from study entry until delivery- anticipated 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Buccal Misoprostol/Vaginal Placebo | Vaginal Misoprostol/Buccal Placebo
Number analyzed (Participants) | 148 | 152
Participants | 14 | 5

3. Secondary Outcome: Number of Vaginal Deliveries That Occurred Within 24 Hours
Description: rate of achieving vaginal delivery within 24 hours
Time Frame: from study entry until delivery- anticipated 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Buccal Misoprostol/Vaginal Placebo | Vaginal Misoprostol/Buccal Placebo
Number analyzed (Participants) | 148 | 152
Participants | 58 | 89

4. Secondary Outcome: Number of Participants Who Had Uterine Hyperstimulation
Description: Presence of uterine hyperstimulation, tachysystole as defined as 6 uterine contractions in a 10 minute period
Time Frame: from study entry until delivery- anticipated 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Buccal Misoprostol/Vaginal Placebo | Vaginal Misoprostol/Buccal Placebo
Number analyzed (Participants) | 148 | 152
Participants | 18 | 22

5. Secondary Outcome: Number of Neonatal Intensive Care Unit (NICU) Admission
Description: Admission to NICU
Time Frame: from study entry until discharge of newborn- anticipated up to 28 days
Measure: Number; unit: participants
Arm/Group | Buccal Misoprostol/Vaginal Placebo | Vaginal Misoprostol/Buccal Placebo
Number analyzed (Participants) | 148 | 152
participants | 30 | 31

6. Secondary Outcome: Number of Doses Misoprostol Used
Description: Number of doses of misoprostol needed
Time Frame: from study entry until delivery- anticipated 3 days
Measure: Median (Full Range); unit: doses
Arm/Group | Buccal Misoprostol/Vaginal Placebo | Vaginal Misoprostol/Buccal Placebo
Number analyzed (Participants) | 148 | 152
doses | 3 [1 to 7] | 2 [1 to 5]

7. Secondary Outcome: Uterine Rupture
Description: Presence of uterine rupture
Time Frame: from study entry until delivery- anticipated 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Buccal Misoprostol/Vaginal Placebo | Vaginal Misoprostol/Buccal Placebo
Number analyzed (Participants) | 148 | 152
Participants | 0 | 0

8. Secondary Outcome: Dose of Oxytocin Used for Augmentation
Description: dose of oxytocin used for augmentation of labor
Time Frame: from study entry until delivery- anticipated 3 days
Measure: Median (Full Range); unit: milliunits per minute
Arm/Group | Buccal Misoprostol/Vaginal Placebo | Vaginal Misoprostol/Buccal Placebo
Number analyzed (Participants) | 148 | 152
milliunits per minute | 6 [0 to 30] | 4 [0 to 36]

9. Secondary Outcome: Number of Participants With Neonatal Cord Gases Measured
Description: cord gases from newborn
Time Frame: from study entry until delivery- anticipated 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Buccal Misoprostol/Vaginal Placebo | Vaginal Misoprostol/Buccal Placebo
Number analyzed (Participants) | 148 | 152
Participants | 12 | 15

10. Other Pre Specified Outcome: Pharmacokinetic Profiling of Misoprostol
Description: pharmacokinetic parameters (Area under the curve, half-life, maximum concentration) measured over first 2 study drug doses
Time Frame: from study entry until delivery- anticipated 3 days
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Participant Satisfaction
Description: participant satisfaction with labor induction and preference for method of drug administration. This will use a questionnaire developed for this study with some similarity to the referenced Nassar study below.
Time Frame: from study entry until discharge- anticipated 5 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Maternal and neonatal adverse events were tracked starting from the first dose and ending at neonatal discharge or thirty days of life, whichever is greater..
Arm/Group | Buccal Misoprostol/Vaginal Placebo | Vaginal Misoprostol/Buccal Placebo
All-Cause Mortality (participants affected / at risk) | 0/148 | 0/152
Serious Adverse Events (participants affected / at risk) | 11/148 | 9/152
Other Adverse Events (participants affected / at risk) | 68/148 | 71/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buccal Misoprostol/Vaginal Placebo (N=148) | Vaginal Misoprostol/Buccal Placebo (N=152)
Inpatient or Postpartum Hospitalization (General disorders) | 11 (11) | 8 (11) — Preeclampsia; Depression; Wound infection; Hemiperitoneum; Endometritis; Herniated disc; Headache; Seizures
Other Life Threatening Event (Pregnancy, puerperium and perinatal conditions) | 0 | 1 (1) — Postpartum hemorrhage
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buccal Misoprostol/Vaginal Placebo (N=148) | Vaginal Misoprostol/Buccal Placebo (N=152)
Any Maternal or Fetal Event (Pregnancy, puerperium and perinatal conditions) | 68 (68) | 71 (71) — allergic reaction to misoprostol; tachysystole requiring therapeutic intervention; cesarean delivery for fetal distress; Appearance, Pulse, Grimace, Activity, Respiration (APGAR) score at 5 minutes less than 7; NICU admission; cord gas pH<7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-12): https://cdn.clinicaltrials.gov/large-docs/15/NCT02408315/Prot_SAP_000.pdf